CLINICAL TRIAL: NCT03136978
Title: Evaluation of Evaluate M1 and M2 Macrophages in Endometriotic Tissue of Women Affected by Endometriosis at Different Stages.
Brief Title: Evaluation of M1 and M2 Macrophages in Endometriotic Tissue of Women Affected by Endometriosis at Different Stages.
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Collaborators: University of Ljubljana (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Messina
Other Study IDs: ENDOMAC
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Endometriosis
Keywords: Macrophages; Macrophages, Peritoneal; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Endometriotic tissue (histologically confirmed) from patients affected by endometriosis at different stages (cases).
  * Tissue samples from ovarian functional cysts (controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: Patients affected by endometriosis (histologically confirmed) at different stages, who will undergo laparoscopic surgery.
  Interventions: Diagnostic Test: Evaluation of M1 and M2 macrophages by flow cytometry.
- Ovarian functional cysts: Patients affected by ovarian functional cysts, who will undergo laparoscopic surgery.
  Interventions: Diagnostic Test: Evaluation of M1 and M2 macrophages by flow cytometry.

INTERVENTIONS:
Diagnostic Test: Evaluation of M1 and M2 macrophages by flow cytometry. — To assess surface expression of macrophage markers, tissue samples will be stained for flow cytometry with fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CCR7 and CD80 to identify M1, whereas fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CD163 and CD206 to identify M2.

SUMMARY:
Accumulating evidence suggests that the peritoneal microenvironment of women affected by endometriosis undergoes a number of local inflammatory-reparative phenomena, with the involvement of resident macrophages, and the attraction and recruitment of peripheral mononuclear cells (monocytes and lymphocytes) from the blood into the peritoneal cavity: during endometriosis a breakdown occurs in endometrial and peritoneal homeostasis caused by cytokine-addressed cell proliferation and dysregulation of apoptosis.

The surrounding microenvironment may address the macrophage plasticity towards a transient and reversible polarization. These polarized phenotypes reflects the proinflammatory or anti-inflammatory status and may change over the time. They could be functionally classified in two main populations: "classically activated" macrophages (M1) and "alternatively activated" macrophages (M2).

Considering that published data so far are still not robust enough to drawn firm conclusion, the aim of this research project will be to evaluate M1 and M2 macrophages in endometriotic tissue from women affected by endometriosis at different stages.

DETAILED DESCRIPTION:
Background and rationale: Endometriosis is an estrogen-dependent disease defined by the ectopic presence and growth of functional endometrial tissue, glands and stroma, outside the uterine cavity (Kavoussi et al, 2016). The aetiopathogenesis of endometriosis still remains controversial: immune, hormonal, genetic, and epigenetic factors may be all involved, and several theories have been proposed to explain it.

The disease affects 2-10 % of women of reproductive age and 50 % of those infertile (Dunselman et al, 2014) and may cause pelvic pain (Triolo et al, 2013; Butticè et al, 2013), abnormal bleeding, infertility/sterility and, consequently, important psychological problems (Laganà et al, 2015). Endometriosis is classified depending on the number, size, and superficial and/or deep location of endometrial implants, plaques, endometriomas and/or adhesions. The most used classification of endometriosis was developed by the American Society for Reproductive Medicine (Rock JA, 1995), although other classification can be used for deep infiltrating endometriosis (Haas et al, 2011) or to correlate endometriosis and infertility (Adamson et al, 2010).

As widely evidenced (Donnez et al, 2016), it is generally accepted that moderate/severe endometriosis-related sterility is due to mechanical factors, namely to the distortion/subversion of the regular pelvic anatomy. On the contrary, the factors behind infertility/subfertility related to minimal/mild endometriosis are less clear. Nevertheless, to date none of the hypothesized mechanisms exhaustively explained the infertility related to endometriosis, while it is possible that such disease is caused by multiple factors altogether, including genetic and epigenetic modifications (Sofo et al, 2015; Maniglio et al, 2016).

Accumulating evidence (Laganà et al, 2013; Laganà et al, 2016) suggests that the peritoneal microenvironment of women affected by endometriosis undergoes a number of local inflammatory-reparative phenomena, with the involvement of resident macrophages, and the attraction and recruitment of peripheral mononuclear cells (monocytes and lymphocytes) from the blood into the peritoneal cavity: during endometriosis a breakdown occurs in endometrial and peritoneal homeostasis caused by cytokine-addressed cell proliferation (Pizzo et al, 2002) and dysregulation of apoptosis (Sturlese et al, 2011; Salmeri et al, 2015).

Monocytes play a key role during adaptive immunity, since they migrates in sites of infection or inflammation, differentiate in macrophages and act as Antigene Presenting Cells (APCs).

Since their first identification of phagocytosis by Elie Metchnikoff in Messina (JAMA, 1968), after experimenting on the larvae of starfish, many steps forward allowed us to have a wide overview of macrophages apart from their role as phagocytic cells.

The surrounding microenvironment may address the macrophage plasticity towards a transient and reversible polarization. These polarized phenotypes reflects the proinflammatory or anti-inflammatory status and may change over the time. They could be functionally classified in two main populations: "classically activated" macrophages (M1) and "alternatively activated" macrophages (M2) (Sica & Mantovani, 2012). Although it is widely accepted that M1 and M2 represent two terminals of the full spectrum of macrophage activation (Liu et al, 2014), recent data (Locati et al, 2013; Mantovani et al, 2013; Capobianco & Rovere-Querini, 2013) allowed to characterize these two populations as follow:

* M1 Macrophages: CD14+ CD68+ CCR7+ CD80+
* M2 Macrophages: CD14+ CD68+ CD163+ CD206+

Study Population: The investigators will select patients affected by histologically confirmed endometriosis (cases) and by ovarian functional cysts (controls), who will undergo laparoscopic surgery. In accordance with the revised American Society for Reproductive Medicine classification for endometriosis (Rock JA, 1995), endometriotic patients will be divided into 4 groups: minimal, mild, moderate and severe stages of endometriosis.

All the laparoscopic procedure will be performed during the proliferative phase of the menstrual cycle. The investigators will exclude from the study women affected by other pelvic disorders, chronic circulatory, autoimmune or neoplastic disease and who took any anti-inflammatory or hormonal or immunomodulatory medication in the preceding 6 months.

Tissue sample preparation and macrophage characterization: Tissue sections (endometriotic tissues for cases, ovarian functional cysts for controls) will be minced and incubated in an enzyme cocktail containing final concentrations of 3.4 mg/ml pancreatin, 0.1 mg/ml hyaluronidase and 1.6 mg/ml collagenase I in Hank's Buffered Saline Solution (HBSS) containing 2 mg/ml D-glucose at 37°C for 2 hours. Following digestion, cells will be dispersed by straining through a 250 μm mesh screen and washed with HBSS. Tissue cells will be stained and fixed for flow cytometric analysis. Prior to macrophage isolation, dead cells will be removed from the culture using the dead cell removal kit. Cell viability will be assessed by trypan blue exclusion.

To assess surface expression of macrophage markers, tissue samples will be stained for flow cytometry with fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CCR7 and CD80 to identify M1, whereas fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CD163 and CD206 to identify M2.

Statistical analysis: The assumption of normal distribution for continuous variables will be tested by Kolmogorov-Smirnov test for goodness of fit. All inferential analyses will be performed using nonparametric statistical tests. Non-normally distributed variables between the groups will be compared using the Kruskal-Wallis test. The range of statistical significance will be P < .05. In addition, The investigators will use post hoc multiple comparison tests either versus controls or versus each stage to analyze data.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by histologically confirmed endometriosis (cases)
* Patients affected by ovarian function cysts (controls)

Exclusion Criteria:

* Other pelvic disorders (apart ovarian functional cysts)
* Chronic circulatory disorders
* Autoimmune disorders
* Neoplastic disorders
* Patients who were treated with any anti-inflammatory or hormonal or immunomodulatory medication in the preceding 6 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients.
Study Population: Reproductive-aged patients affected by histologically confirmed endometriosis (cases) and by ovarian functional cysts (controls), who will undergo laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Quantification of M1 and M2 macrophages in endometriotic tissue for each stage of endometriosis. | Day 1
  To assess surface expression of macrophage markers, endometrial tissue cells will be stained for flow cytometry with fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CCR7 and CD80 to identify M1, whereas fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CD163 and CD206 to identify M2.

SECONDARY OUTCOMES:
Correlation of M1 and M2 macrophages quantity in endometriotic tissue to the presence of endometriosis-associated infertility. | Day 1
  To assess surface expression of macrophage markers, endometrial tissue cells will be stained for flow cytometry with fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CCR7 and CD80 to identify M1, whereas fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CD163 and CD206 to identify M2. Female infertility will be defined by the failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse.
Correlation of M1 and M2 macrophages quantity in endometriotic tissue to the presence of endometriosis-associated chronic pelvic pain. | Day 1
  To assess surface expression of macrophage markers, endometrial tissue cells will be stained for flow cytometry with fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CCR7 and CD80 to identify M1, whereas fluorochrome-conjugated monoclonal antibodies against CD14, CD68, CD163 and CD206 to identify M2. Chronic pelvic pain will be defined as pain that occurs below the umbilicus (belly button) that lasts for at least six months.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kavoussi SK, Lim CS, Skinner BD, Lebovic DI, As-Sanie S. New paradigms in the diagnosis and management of endometriosis. Curr Opin Obstet Gynecol. 2016 Aug;28(4):267-76. doi: 10.1097/GCO.0000000000000288. PMID 27306924
- [Background] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Background] Triolo O, Lagana AS, Sturlese E. Chronic pelvic pain in endometriosis: an overview. J Clin Med Res. 2013 Jun;5(3):153-63. doi: 10.4021/jocmr1288w. Epub 2013 Apr 23. PMID 23671540
- [Background] Buttice S, Lagana AS, Barresi V, Inferrera A, Mucciardi G, Di Benedetto A, D'Amico CE, Magno C. Lumbar Ureteral Stenosis due to Endometriosis: Our Experience and Review of the Literature. Case Rep Urol. 2013;2013:812475. doi: 10.1155/2013/812475. Epub 2013 May 2. PMID 23738189
- [Background] Lagana AS, Condemi I, Retto G, Muscatello MR, Bruno A, Zoccali RA, Triolo O, Cedro C. Analysis of psychopathological comorbidity behind the common symptoms and signs of endometriosis. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:30-3. doi: 10.1016/j.ejogrb.2015.08.015. Epub 2015 Aug 15. PMID 26319653
- [Background] Rock JA. The revised American Fertility Society classification of endometriosis: reproducibility of scoring. ZOLADEX Endometriosis Study Group. Fertil Steril. 1995 May;63(5):1108-10. doi: 10.1016/s0015-0282(16)57556-6. PMID 7720925
- [Background] Haas D, Chvatal R, Habelsberger A, Wurm P, Schimetta W, Oppelt P. Comparison of revised American Fertility Society and ENZIAN staging: a critical evaluation of classifications of endometriosis on the basis of our patient population. Fertil Steril. 2011 Apr;95(5):1574-8. doi: 10.1016/j.fertnstert.2011.01.135. PMID 21315335
- [Background] Adamson GD, Pasta DJ. Endometriosis fertility index: the new, validated endometriosis staging system. Fertil Steril. 2010 Oct;94(5):1609-15. doi: 10.1016/j.fertnstert.2009.09.035. PMID 19931076
- [Background] Donnez J, Donnez O, Orellana R, Binda MM, Dolmans MM. Endometriosis and infertility. Panminerva Med. 2016 Jun;58(2):143-50. Epub 2016 Feb 2. PMID 26837776
- [Background] Sofo V, Gotte M, Lagana AS, Salmeri FM, Triolo O, Sturlese E, Retto G, Alfa M, Granese R, Abrao MS. Correlation between dioxin and endometriosis: an epigenetic route to unravel the pathogenesis of the disease. Arch Gynecol Obstet. 2015 Nov;292(5):973-86. doi: 10.1007/s00404-015-3739-5. Epub 2015 Apr 29. PMID 25920525
- [Background] Maniglio P, Ricciardi E, Lagana AS, Triolo O, Caserta D. Epigenetic modifications of primordial reproductive tract: A common etiologic pathway for Mayer-Rokitansky-Kuster-Hauser Syndrome and endometriosis? Med Hypotheses. 2016 May;90:4-5. doi: 10.1016/j.mehy.2016.02.015. Epub 2016 Feb 27. No abstract available. PMID 27063075
- [Background] Lagana AS, Sturlese E, Retto G, Sofo V, Triolo O. Interplay between Misplaced Mullerian-Derived Stem Cells and Peritoneal Immune Dysregulation in the Pathogenesis of Endometriosis. Obstet Gynecol Int. 2013;2013:527041. doi: 10.1155/2013/527041. Epub 2013 Jun 13. PMID 23843796
- [Background] Lagana AS, Triolo O, Salmeri FM, Granese R, Palmara VI, Ban Frangez H, Vrtcnik Bokal E, Sofo V. Natural Killer T cell subsets in eutopic and ectopic endometrium: a fresh look to a busy corner. Arch Gynecol Obstet. 2016 May;293(5):941-9. doi: 10.1007/s00404-015-4004-7. Epub 2016 Jan 6. PMID 26739265
- [Background] Pizzo A, Salmeri FM, Ardita FV, Sofo V, Tripepi M, Marsico S. Behaviour of cytokine levels in serum and peritoneal fluid of women with endometriosis. Gynecol Obstet Invest. 2002;54(2):82-7. doi: 10.1159/000067717. PMID 12566749
- [Background] Sturlese E, Salmeri FM, Retto G, Pizzo A, De Dominici R, Ardita FV, Borrielli I, Licata N, Lagana AS, Sofo V. Dysregulation of the Fas/FasL system in mononuclear cells recovered from peritoneal fluid of women with endometriosis. J Reprod Immunol. 2011 Dec;92(1-2):74-81. doi: 10.1016/j.jri.2011.08.005. Epub 2011 Oct 5. PMID 21978769
- [Background] Salmeri FM, Lagana AS, Sofo V, Triolo O, Sturlese E, Retto G, Pizzo A, D'Ascola A, Campo S. Behavior of tumor necrosis factor-alpha and tumor necrosis factor receptor 1/tumor necrosis factor receptor 2 system in mononuclear cells recovered from peritoneal fluid of women with endometriosis at different stages. Reprod Sci. 2015 Feb;22(2):165-72. doi: 10.1177/1933719114536472. Epub 2014 May 20. PMID 24844917
- [Background] Elie Metchnikoff (1845-1916), advocate of phagocytosis. JAMA. 1968 Jan 8;203(2):139-41. No abstract available. PMID 4864332
- [Background] Sica A, Mantovani A. Macrophage plasticity and polarization: in vivo veritas. J Clin Invest. 2012 Mar;122(3):787-95. doi: 10.1172/JCI59643. Epub 2012 Mar 1. PMID 22378047
- [Background] Liu YC, Zou XB, Chai YF, Yao YM. Macrophage polarization in inflammatory diseases. Int J Biol Sci. 2014 May 1;10(5):520-9. doi: 10.7150/ijbs.8879. eCollection 2014. PMID 24910531
- [Background] Locati M, Mantovani A, Sica A. Macrophage activation and polarization as an adaptive component of innate immunity. Adv Immunol. 2013;120:163-84. doi: 10.1016/B978-0-12-417028-5.00006-5. PMID 24070384
- [Background] Mantovani A, Biswas SK, Galdiero MR, Sica A, Locati M. Macrophage plasticity and polarization in tissue repair and remodelling. J Pathol. 2013 Jan;229(2):176-85. doi: 10.1002/path.4133. Epub 2012 Nov 29. PMID 23096265
- [Background] Capobianco A, Rovere-Querini P. Endometriosis, a disease of the macrophage. Front Immunol. 2013 Jan 28;4:9. doi: 10.3389/fimmu.2013.00009. eCollection 2013. PMID 23372570